CLINICAL TRIAL: NCT00326274
Title: Clinical Safety Trial of Long-Term Intermittent Use of Helioblock® SX Cream
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Loreal USA (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: PEN.750.04
Record Dates: First submitted 2006-05-15; First posted 2006-05-16 (Estimated); Last update posted 2009-02-11 (Estimated); Status verified 2009-02

CONDITIONS: Sunburn
MeSH Terms: conditions — Sunburn

INTERVENTIONS:
Drug: Helioblock® SX Cream

SUMMARY:
The purpose of this study is to determine the safety potential of Helioblock® SX Cream as a sunscreen product in long term intermittent use conditions among pediatric subjects.. Each subject will be enrolled to participate for six months. The test product should be applied every day that outdoor activities are planned, prior to any significant sun exposure during out-door activities (such as the beach, outdoor sport activities), or whenever the subject needs to be protected against sunburn or other damage due to the sun. A minimum of 14 days test product use and sun exposure is required.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects of any race or skin type, 6 months to 12 years of age inclusive, willing to use the test product intermittently for six months during outside activities

Exclusion Criteria:

* Subjects with known sensitivities to any of the study ingredients or subjects with a condition or in a situation, which in the Investigator's opinion, may suggest a significant hazard for the subject, may confound the study results, or interfere with the subject's participation in the study.
* Subjects who are pregnant or lactating

Ages: 6 Months to 12 Years | Sex: All
Age Groups: Child
Dates: Start 2006-05; Primary Completion 2006-11 (Actual); Study Completion 2006-11

PRIMARY OUTCOMES:
Long term safety after 6 months intermittent use in a pediatric population | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Research Testing Laboratories, Great Neck, New York, United States